CLINICAL TRIAL: NCT02805205
Title: A Multi-center, Open-label,Single Arm Phase IV Clinical Trial of Efficacy and Safety of PEG-rhG-CSF in Preventing Neutropenia in Patients With Breast Cancer Receiving Chemotherapy
Brief Title: PEG-rhG-CSF in Patients With Breast Cancer Receiving Chemotherapy to Prevent Neutropenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: CSPC Baike (Shandong) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CSPC-PGC-IV-02
Record Dates: First submitted 2016-06-13; First posted 2016-06-17 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
Keywords: PEG-rhG-CSF neutropenia
MeSH Terms: conditions — Breast Neoplasms | interventions — pegylated granulocyte colony-stimulating factor; pegfilgrastim

ARMS (1):
- PEG-rhG-CSF (Experimental): patients received a single dose of 100 ug/kg of PEG-rhG-CSF(pegfilgrastim), on the basis of actual body weight, as a single subcutaneous injection on day 3 after chemotherapy
  Interventions: Drug: PEG-rhG-CSF

INTERVENTIONS:
Drug: PEG-rhG-CSF
  Other Names: pegfilgrastim

SUMMARY:
The purpose of this study is to estimate the efficacy and safety of PEG-rhG-CSF in patients with breast cancer receiving chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age between 18 and 70 years
* diagnosis of breast cancer patients who need to receive multi-cycle chemotherapy
* grade III/IV neutropenia after chemotherapy
* KPS score≥70
* life expectancy of at least 3 months
* Written informed consent are acquired

Exclusion Criteria:

* Have accepted any other drug related clinical trial within 4 weeks before anticipated
* uncontrolled infection
* pregnancy
* Other situations that investigators consider as contra-indication for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2013-04; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
the occurrence rate of the adverse events that are related to treatment during four consecutive cycles chemotherapy | up to 30 days after the patient study completion
the severity of the adverse events that are related to treatment during four consecutive cycles chemotherapy | up to 30 days after the patient study completion

SECONDARY OUTCOMES:
the occurrence rate of III/ IV neutropenia during the whole chemotherapy process | through the study completion,an average of 5 months